CLINICAL TRIAL: NCT07012044
Title: A Phase 1 Study of Oral Cedazuridine and Decitabine Combination (ASTX727, NSC# 820631) and Filgrastim as Maintenance Therapy Post-Hematopoietic Stem Cell Transplant in Children With High-Risk Acute Myeloid Leukemia
Brief Title: A Study to Find the Highest Dose of Cedazuridine and Decitabine Combination With Filgrastim as a Treatment Option After Hematopoietic Stem Cell Transplant in Children With High-Risk Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-03946; NCI-2025-03946 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEPN2413 (Other: Pediatric Early Phase Clinical Trial Network); PEPN2413 (Other: CTEP); UM1CA228823 (NIH)
Record Dates: First submitted 2025-06-07; First posted 2025-06-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia Post Cytotoxic Therapy; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; Decitabine; Injections; decitabine and cedazuridine drug combination; Filgrastim; Granulocyte Colony-Stimulating Factor; X-Rays; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ASTX727, diecitabine, filgrastim) (Experimental): Patients receive filgrastim SC or IV QD on days 1-6 and ASTX727 PO QD on days 2-6. Patients may receive decitabine PO QD on days 2-6 to achieve the appropriate dose. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy and blood sample collection throughout the study and may undergo lumbar puncture and diagnostic imaging throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine; Drug: Decitabine and Cedazuridine; Biological: Filgrastim; Procedure: Imaging Procedure; Procedure: Lumbar Puncture

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Decitabine — Given PO
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Biological: Filgrastim — Given SC or IV
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Procedure: Imaging Procedure — Undergo diagnostic imaging
  Other Names: Diagnostic Imaging Technique; Image Type; Imaging; Imaging (procedure); Imaging Procedures; Imaging Technique; imaging type; IMAGING_METHOD; imaging_type; Medical Imaging; Type of imaging
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of ASTX727 and filgrastim for the treatment of children with high risk acute myeloid leukemia that has come back after a period of improvement (recurrent) or that does not respond to treatment (refractory) who have undergone allogenic hematopoietic stem cell transplantation. ASTX727 is a combination of cedazuridine and decitabine. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Filgrastim stimulates the production of neutrophils (a type of white blood cell) which can help to prevent infection. Giving ATSX727 and filgrastim may be safe and tolerable in treating children with high risk, recurrent or refractory acute myeloid leukemia who have undergone allogenic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose and/or recommended phase 2 dose (RP2D) of decitabine and cedazuridine (ASTX727) administered together with filgrastim (rh-granulocyte colony stimulating factor [GCSF]) post-hematopoietic stem cell transplant (HCT) to children with high-risk acute myeloid leukemia (AML).

II. To define and describe the toxicities of ASTX727 administered together with filgrastim (rh-GCSF) post-HCT in children with high-risk AML.

III. To characterize the pharmacokinetic profile of ASTX727 administered together with filgrastim (rh-GCSF) post-HCT in children with high-risk AML.

SECONDARY OBJECTIVES:

I. To determine the incidence and severity of graft versus host disease and graft rejection in children with high-risk AML who received post-HCT therapy with ASTX727 and filgrastim (rh-GCSF).

II. To preliminarily describe the 1-year event free survival (EFS) of patients with AML who received post-HCT therapy with ASTX727 and filgrastim (rh-GCSF), within the confines of a phase 1 study.

EXPLORATORY OBJECTIVE:

I. To characterize the pharmacodynamic profile of ASTX727 through deoxyribonucleic acid (DNA) methylation assay and, in turn, the potential impact of hypomethylation on donor immune cells and the graft versus leukemia effect.

OUTLINE: This is a dose-escalation study of decitabine in combination with cedazuridine and filgrastim.

Patients receive filgrastim subcutaneously (SC) or intravenously (IV) once daily (QD) on days 1-6 and ASTX727 orally (PO) QD on days 2-6. Patients may receive decitabine PO QD on days 2-6 to achieve the appropriate dose. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy and blood sample collection throughout the study and may undergo lumbar puncture and diagnostic imaging throughout the study.

After completion of study treatment, patients are followed up at 1 year post transplant and/or at relapse.

ELIGIBILITY:
Inclusion Criteria:

* STEP 0: Patient must be ≤ 21 years of age

  * PLEASE NOTE: Eligibility criteria to enroll onto Step 1 for the treatment trial is ≤ 21 years of age at the time of Step 1 enrollment. Please plan accordingly to ensure that patients who are screened with Step 0 will be at an eligible age at the time of enrollment onto Step 1. Patients who are 21 at the time of screening who turn 22 at the time of enrollment onto Step 1 will not be eligible to enroll onto the study
* STEP 0: Patients with newly diagnosed high risk* de novo AML, newly diagnosed therapy-related AML, relapsed, or refractory AML. Patients with isolated or combined central nervous system (CNS) or extramedullary disease are eligible

  * Based on risk criteria adopted by the AAML1831 study
* STEP 0: Patient must plan to have bone marrow sample submitted to Hematologics within 14 days prior to the start of conditioning regimen for HCT.

  * Note: In order to be eligible to enroll onto Step 1 to receive treatment on this study, pre-HCT disease status must be assessed prior to receiving HCT. AML must be in complete remission (Children's Oncology Group [COG]-complete remission [CR], COG-complete remission with partial recovery of platelelt count [CRp], COG-complete remission with incomplete blood count recovery [Cri], with or without detectable minimal residual disease [MRD]); bone marrow CR must be assessed by central flow cytometry performed at Hematologics prior to receiving HCT
* STEP 0: Human immunodeficiency virus (HIV)-infected patients are eligible for this trial if the following criteria are met:

  * No history of HIV complications with the exception of CD4 count < 200cells/mm^3
  * No antiretroviral therapy with overlapping toxicity such as myelosuppression
  * CD4 count > 500 cells/mm^3 prior to the diagnosis of newly diagnosed, relapsed, refractory AML.
  * HIV viral loads below the limit of detection within 6 months, as long as the patient is NOT receiving anti-retroviral agents that may interact with ASTX727.
  * No history of highly active antiretroviral therapy (HAART)-resistant HIV
* STEP 0: Patients must be receiving an allogeneic (related, unrelated, and mismatched related, including haploidentical) marrow, peripheral blood, or cord blood transplant for the first time
* STEP 0: HCT conditioning regimen must be planned to begin within 14 days after bone marrow MRD assessment to determine disease status
* STEP 0: Conditioning regimen must be myeloablative and include high dose busulfan, or treosulfan, or total body irradiation
* STEP 0: Patients must not have received prior exposure to ASTX727. Note that patients may have had prior exposure to decitabine
* STEP 1: Patient must be ≤ 21 years of age at the time of study enrollment to step 0
* STEP 1: Patients must have a body surface area ≥ 1m^2 at enrollment to step 1
* STEP 1 (PRE-HCT): AML must be in complete remission (COG-CR, COG-CRp, COG-Cri, with or without detectable MRD); bone marrow CR must be assessed by central flow cytometry performed at Hematologics. Disease assessment must be performed within 14 days prior to HCT conditioning regimen
* STEP 1 (POST-HCT): AML must be in complete remission (COG-CR, COG-CRp, COG-CRi). Bone marrow evaluation must show CR with no detectable minimal residual disease (MRD negative by central flow cytometry at Hematologics)

  * Note: Disease assessment is required to be performed within 14 days prior to enrollment onto Step 1
* STEP 1: Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age. Patients must have Karnofsky performance score ≥ 50 or Lansky play-performance scale score ≥ 50
* STEP 1: Patients must have fully recovered from the acute toxicities related to the conditioning regimen and the transplant. If, after 42-100 days post-transplant, the eligibility criteria are met, the patient is considered to have recovered adequately
* STEP 1: Platelet count ≥ 20,000 µL (without requirement for platelet transfusion within the last 7 days)
* STEP 1: Hemoglobin ≥ 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions)
* STEP 1: Absolute neutrophil count ≥ 1,000 µL with no myeloid growth factor support within the last 3 days
* STEP 1:

  * 1 month to < 6 months: Maximum serum creatinine 0.4 mg/dL (male), 0.4 mg/dL (female)
  * 6 months to < 1 year: Maximum serum creatinine 0.5 mg/dL (male), 0.6 mg/dL (female)
  * 1 to < 2 years: Maximum serum creatinine 0.6 mg/dL (male), 0.6 mg/dL (female)
  * 2 to < 6 years: Maximum serum creatinine 0.8 mg/dL (male), 0.8 mg/dL (female)
  * 6 to < 10 years: Maximum serum creatinine 1 mg/dL (male), 1 mg/dL (female)
  * 10 to < 13 years: Maximum serum creatinine 1.2 mg/dL (male), 1.2 mg/dL (female)
  * 13 to < 16 years: Maximum serum creatinine 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years: Maximum serum creatinine 1.7 mg/dL (male),1.4 mg/dL (female) OR a 24 hour urine creatinine clearance ≥ 60 mL/min/1.73 m^2 OR a glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard).
  * Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility
* STEP 1: Bilirubin (total or sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
* STEP 1: Alanine aminotransferase (ALT) ≤ 3 x ULN, unless attributed to leukemia or tumor involvement then ALT ≤ 5 x ULN
* STEP 1: Aspartate aminotransferase (AST) ≤ 3 x ULN, unless attributed to leukemia or tumor involvement then AST ≤ 5 x ULN
* STEP 1: Albumin ≥ 2 g/dL

Exclusion Criteria:

* STEP 0: Patients with known inherited marrow failure syndromes, including, but not limited to Fanconi Anemia, Dyskeratosis congenita, and Shwachman-Diamond syndrome
* STEP 0: Known or suspected hypersensitivity to filgrastim, decitabine or cedazuridine (ASTX727)
* STEP 0: Patients who have received a prior solid organ transplantation are not eligible
* STEP 1: ASTX727 can cause fetal harm when administered to pregnant women. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method (eg, male or female condom) for the duration of the study. Abstinence is an acceptable method of birth control. Women of childbearing potential must use highly effective contraception during treatment with ASTX727 and for at least 6 months after the last dose. Men with female partners of childbearing potential should be advised to practice highly effective contraceptive measures of birth control and not to father a child while receiving treatment with decitabine and for 3 months after the last dose. Breastfeeding is not allowed during the study and for at least 2 weeks after the last dose of study drug
* STEP 1: Patients who are currently receiving another investigational drug are not eligible
* STEP 1: Patients who are currently receiving other anti-cancer agents are not eligible
* STEP 1: Patients receiving or for whom there is a plan to administer anticancer directed non-protocol therapy, radiation therapy or immunotherapy during the study period are not eligible (note that prophylactic use of chemotherapeutic agents for graft versus host disease [GVHD] is allowed, e.g. methotrexate for GVHD prophylaxis). Intrathecal chemotherapy administered at the discretion of the treating physician throughout maintenance therapy is allowed
* STEP 1: Drugs known to be metabolized by cytidine deaminase (CDA) should not be given (such drugs include cytarabine, gemcitabine, azacitidine, vidarabine, zalcitabine, zidovudine, telbivudine, didanosine, stavudine, lamivudine, abacavir, emtricitabine, entecavir, trifluridine, tenofovir and adefovir) on days when ASTX727 is administered and for 24 hours thereafter
* STEP 1: Patients is not able to swallow intact tablets. Nasogastric or G tube administration is not allowed
* STEP 1: Patient is not able to start ASTX727 and filgrastim (rh-GCSF) between day 42 and day 100 following completion of allo-HCT. If, after enrollment, protocol therapy is started more than 60 days following allo-HCT, the patient will be removed from protocol therapy
* STEP 1: Patients with graft loss are not eligible
* STEP 1: Patients with steroid refractory or dependent acute GVHD are not eligible. Patients must be on < 1 mg/kg/day of methylprednisolone (or equivalent prednisone/prednisolone dose) that is being tapered. Patients must not be on any second line systemic therapies. Continued GVHD prophylaxis with calcineurin inhibitors, sirolimus, abatacept or mycophenolate mofetil is acceptable
* STEP 1: Patients who have an uncontrolled viral, bacterial, fungal, or protozoal infection are not eligible
* STEP 1: Patients with active transplant associated thrombotic microangiopathy with ongoing hemolysis and need treatment (e.g. eculizumab) are not eligible
* STEP 1: Patients with sinusoidal obstruction syndrome with ongoing need for treatment (e.g. defibrotide, diuresis, supplemental oxygen) are not eligible
* STEP 1: Idiopathic pneumonitis syndrome or other non-infectious lung injury requiring ongoing treatment (corticosteroids, tumor necrosis factor [TNF] inhibitors, or other biologics) or supplemental oxygen are not eligible
* STEP 1: Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-04-29 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to completion of cycle 2 (cycle length=28 days)
  Defined as maximum dose at which fewer than one-third of patients experience dose limiting toxicity.
Incidence of adverse events | Up to 2 years
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Pharmacokinetic profile of ASTX727 | At cycle 1 last day of dosing
  Will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).

SECONDARY OUTCOMES:
Incidence of graft versus host disease | Up to 2 years
Severity of graft versus host disease | Up to 2 years
Incidence of graft rejection | Up to 2 years
Severity of graft rejection | Up to 2 years
Event free survival | At 1 year

OTHER OUTCOMES:
Pharmacodynamic profile of ASTX727 | At cycle 1 day 1 and cycle 1 day 8
  Assessed through deoxyribonucleic acid methylation assay.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Sulis, Principal Investigator — Pediatric Early Phase Clinical Trial Network

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm